CLINICAL TRIAL: NCT00193804
Title: A Phase II Randomized Trial Comparing Intensity Modulated Radiation Therapy (IMRT) With Conventional Radiation Therapy in Stage IIB Carcinoma Cervix
Brief Title: A Trial Comparing Intensity Modulated Radiation Therapy (IMRT) With Conventional Radiation Therapy in Stage IIB Carcinoma Cervix
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Sk Shrivastava, Prof. & Head of Radiation Oncology, Tata Memorial Hospital
Other Study IDs: TMH/158/2004/Cx_IMRT TRIAL
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Cancer of Cervix
Keywords: Cervical Cancer; FIGO STAGE IIB; CHEMORADIATION; Intensity Modulated Radiation Therapy(IMRT); Conventional Radiation Therapy; Cancer of the Cervix; Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 2: Patients with histologically proven, cervical cancer FIGO Stage IIB eligible will be invited for the study. The patients will recieve either 3D conformal radiation or IMRT external radiation with concomitant cisplatin chemotherapy followed by brachytherapy.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT — IMRT in cervical cancers

SUMMARY:
A study to evaluate the efficacy of Intensity Modulated Radiation Therapy (IMRT) as compared to Standard Conventional Radiotherapy Alone in the treatment of carcinoma cervix. Concomitant Weekly Cisplatin chemotherapy will be given as a routine, which is a standard of care today for early stage cervical cancers including stage IIB. The benefits of using IMRT in reducing radiation-induced toxicity are well known. Since this treatment modality has not yet been validated and studied in a randomized trial setting, the present study is being undertaken. The study arm of IMRT has the potential to reduce the toxicities by 15-20%, but is associated with labor intense procedure requiring many hospital visits before actual start of treatment.

DETAILED DESCRIPTION:
Carcinoma Cervix is the commonest malignancy seen in Indian women and constitutes approximately 10% of all cancers at Tata Memorial Hospital (1). It is also the leading cause of cancer mortality in India. Nearly 85% of the patients present with advanced stages (FIGO Stage II/III). The main stay of treatment has traditionally been radical radiation therapy with 80-90% of patients requiring radiation in their lifetime and over decades the survival rates have achieved a plateau of 30 - 55% at 5 years.

Radiation therapy is usually a combination of external beam and intracavitary brachytherapy. External beam radiation includes irradiation of primary tumor and nodal areas of risk. Higher Doses of external beam radiation is limited due to normal critical organs namely, small bowel, rectum and bladder. A major concern with pelvic radiation is the considerable volume of both small bowel and rectum is included in the radiation treatment fields. Unsurprisingly, gastrointestinal radiation reactions include diarrhea while late sequelae include small bowel obstruction, enteritis and diarrhea are common (2-4). The benefits of multiple fields, high energy beams, customized blocking and low fraction sizes are well known (4). Various methods have been used to reduce the small bowel complications. Surgical methods include absorbable meshes (5), tissue expanders (6) and omentoplasty (7). However, these approaches are not feasible in patients undergoing definitive radiation. Apart from small bowel toxicity, late rectal and bladder complications are also of a major concern. The clinical manifestations vary from mild proctitis, stricture, bleeding ulcers and fistula formation to hemorrhagic cystitis requiring cystectomy. Grade III radiation cystitis and proctitis reported are in the range of 3-15% with radiation alone.

Moreover, of late the pattern of practice is increasingly being emphasized on concomitant chemo radiation (8,9). The addition of chemotherapy though has no doubt improved the survivals, but has also led to increase in normal tissue toxicities. In the RTOG 90-01 and 92-10 there is alarming increase in the gastro intestinal (35% grade III and grade IV) and genitourinary (9% grade III and grade IV).

The changes in the treatment policies and the toxicities associated with wide pelvic radiation therapy demand for better normal tissue sparing radiation techniques or radioprotective agents. Three Dimensional Conformal Radiation Therapy (3D-CRT) to some extent has successfully achieved some normal tissue sparing. Intensity-modulated radiotherapy (IMRT) is an important recent advance in radiation therapy and is at the forefront of Translational Research. With 3DCRT the radiation intensity is generally uniform within the radiation portal whereas in IMRT the dose intensity within the portal varies with the use of beamlets, thereby allows a higher degree of conformation to the tumor than previously possible and allows concave isodose profiles to be generated.

Over last 10 years, IMRT has been successfully used in the treatment of prostate, head and neck and brain tumors. IMRT in pelvic radiation has the potential to reduce the dose as well as the volume of rectum, bladder and small bowel irradiated significantly and thereby translating into a decrease in the incidence and severity, of acute and late gastro-intestinal and genito-urinary toxicities. Several dosimetric studies have been reported to confirm the role of IMRT in reducing toxicities with pelvic radiation therapy (10,11). These dosimetric studies have reported that the volume of small bowel irradiated to the prescription dose by a factor of 2 compared with conventional radiation. The average volume of bladder and rectum irradiated is also reduced by 23% (12). In our series of 10 patients treated, IMRT in pelvic radiation therapy apart from reducing the hot spot volumes and better conformity index to the target volume, also significantly reduces the volumes of high dose regions in small bowel region (by 17%), rectum (by 50-60%) and bladder (by 40-50%) [unpublished data]. In another series of early report on outcome of 40 patients treated with IMRT to whole pelvis, Arno el al. have demonstrated that there is a significant reduction in acute radiation related toxicities, but it is too early to comment on late sequelae since the follow-up is short and has concluded that, this novel approach definitely needs to be validated in a trial setting. (13)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous carcinoma or adenocarcinoma of cervix
* Performance index WHO grade 0 or 1
* Patients below 65 years of age
* FIGO Stage IIB
* Normal ECG and Cardiovascular system
* Normal hematological parameters
* Normal renal and liver function tests

Exclusion Criteria:

* Co-morbid conditions like medical renal disease
* Medical or Psychological condition that would preclude treatment
* H/o Previous treatment / Pregnancy
* Patient unreliable for treatment completion and follow-up.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven cervical cancers, FIGO Stage IIb eligible for the study will be invited for the study
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-02; Primary Completion 2017-06-20 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
To compare the normal tissue toxicities (Acute & Late) of standard radiation therapy with IMRT | 2017

SECONDARY OUTCOMES:
To compare the disease free survivals | 2017
To compare the quality of life in both the groups | 2017
To compare the overall survivals | 2017

CONTACTS AND LOCATIONS:
Overall Officials: Shyamkishore J Shrivastava, MD, DNB (RT), Principal Investigator — Professor & Head, Radiation Oncology, Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Tata Memorial Hospital — https://tmc.gov.in/